CLINICAL TRIAL: NCT02903329
Title: Efficacy of Restricted Acute Medication Intake Compared to no Acute Medication Intake During a Two Months Detoxification Period in Medication-overuse Headache
Brief Title: Comparison of Two Detoxification Protocols for Treatment of Medication-overuse Headache
Acronym: MUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Louise Carlsen, MD; PhD-student, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1-2012-116
Record Dates: First submitted 2016-09-01; First posted 2016-09-16 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Medication-overuse Headache
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Inactivation, Metabolic; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol A (Active Comparator): In program A, patients underwent detoxification without any acute medication during a two months period (complete stop of acute medication intake).
  Interventions: Other: Detoxification
- Protocol B (Active Comparator): In program B, patients were allowed to take up to 2 days a week with analgesics or migraine medication during the two months detoxification period (restricted acute medication intake).
  Interventions: Other: Detoxification

INTERVENTIONS:
Other: Detoxification — Two ways of composing the detoxification protocol
  Other Names: Treatment for MOH

SUMMARY:
Medication-overuse headache (MOH) is a common, costly and disabling disorder affecting approximately 63 million people worldwide. MOH is a potentially treatable condition, and there are different opinions among headache specialists concerning the correct treatment strategy.

The study is a prospective longitudinal open-label randomized controlled study comparing two detoxification programs conducted in a tertiary headache care center. Patients with MOH are either randomized to treatment in program A or program B. In program A, patients undergo detoxification without any acute medication during a two months period (complete stop of acute medication intake). In program B, patients was allowed to take up to 2 days a week with analgesics or migraine medication during the two months detoxification period (restricted acute medication intake). Both A and B are out-patient programs, and patients in both groups receive patient education, consisting of six lessons, managed by specialized headache nurses in collaboration with specialized psychologists and physiotherapists (Figure 1). All patients are also offered rescue medication (levomepromazine or promethazine) and antiemetics, if necessary.

The need for prophylactic treatment is evaluated individually after 2-month detoxification. Patients are followed-up at 2, 6 and 12 months after detoxification. All patients are asked to continuously register headache calendar and to fulfill questionnaires at all the follow-up visits. In addition they are asked to fill out questionnaires (Headache Under-Response to Treatment (HURT), Hospital Anxiety and Depression Score (HADS), Severity of Dependence Score (SDS), World Health Organization Quality of Life Score(WHO QoL) and Dolo-score) at baseline, 2, 6 and 12 months

DETAILED DESCRIPTION:
Patients with contact to Danish headache center are recruited consecutively. The MOH-diagnosis is based on least 3 months previous detailed history and at least 1 month fulfilled headache diary or headache calendar prior to the visit.

Patients were allocated to either program A or B by a concealed randomization process. The patients were randomized in blocks of 10 by use of opaque, sealed envelopes.

Statistics Statistical Package for Social Sciences (SPSS) version 22 is used for statistical calculations. Continuous variables are presented as mean (SD) and median (25-75 percentiles). For normal distributed continuous variables the investigators use paired and unpaired student's T-test, while for skewed distribution the investigators used Mann-Whitney test. Categorical variables is presented as percentage (N), and analyzed by chi-square test. All results are shown as intention-to-treat (ITT). The p-value is two-sided and p ≤ 0.05 is considered as significant.

The primary outcome is reduction in headache days per month. Clinical relevant difference is estimated to 20% between the two groups. The standard deviation based on previous published literature was estimated to 35%. Accepting an alfa-error on 5% and 80% power, 80 patients are needed. Based on previous studies, it is assumed that the drop-out rate will be approximately 15-20%. Therefore the investigators aim to include 100 patients corresponding to 50 in each group.

ELIGIBILITY:
Inclusion Criteria:

* MOH-diagnosis according to ICHD-3beta
* Eligible for out-patient care
* Previously diagnosed with primary headache forms.

Exclusion Criteria:

* Previously diagnosed with secondary headache forms
* Significant physical or psychiatric illness
* Pregnancy or breastfeeding
* Inadequate language skills to follow the patient education and filling out questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Headache frequency | 6 months

SECONDARY OUTCOMES:
Days with acute medication/ month | 6 and 12 month
Headache frequency | 12 months
Headache intensity (Total intensity per month meassured by headache calendars). | 6 and 12 months
  Patients daily register headache intensity by 0,1, 2 or 3 corresponding to the intensity. The headache intensity is summed up for 30 days.
Scores from questionnaires Headache Under-Response to Treatment (HURT) | 6 and 12 months
Scores from questionnaires Hospital Anxiety and Depression Score (HADS) | 6 and 12 months
Scores from questionnaires World Health Organization Quality of Life score | 6 and 12 months
Scores from questionnaires Severity of Dependence Score (SDS) | 6 and 12 months
Scores from questionnaires Dolo-score | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Louise Ninett Carlsen, MD, Study Chair — Danich Headache Center, Neurological department, Rigshospitalet-Glostrup
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen M, Carlsen LN, Munksgaard SB, Engelstoft IMS, Jensen RH, Bendtsen L. Complete withdrawal is the most effective approach to reduce disability in patients with medication-overuse headache: A randomized controlled open-label trial. Cephalalgia. 2019 Jun;39(7):863-872. doi: 10.1177/0333102419828994. Epub 2019 Feb 7. PMID 30732459
- [Derived] Carlsen LN, Munksgaard SB, Jensen RH, Bendtsen L. Complete detoxification is the most effective treatment of medication-overuse headache: A randomized controlled open-label trial. Cephalalgia. 2018 Feb;38(2):225-236. doi: 10.1177/0333102417737779. Epub 2017 Oct 19. PMID 29050498